CLINICAL TRIAL: NCT03778580
Title: Advanced Glycation Endproducts and Bone Material Strength in Type 2 Diabetes Treated With Pyridoxamine
Brief Title: Advanced Glycation Endproducts and Bone Material Strength in T2D Treated With Pyridoxamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Mishaela Rubin, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAR5451
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vitamin B6; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — pyridoxamine dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pyridoxamine (Experimental): pyridoxamine dihydrochloride (over- the- counter type of vitamin B6) 200 mg po bid for one year
  Interventions: Dietary Supplement: Pyridoxamine Dihydrochloride
- identical placebo (Placebo Comparator): identical placebo po bid for one year
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: Pyridoxamine Dihydrochloride — pyridoxamine dihydrochloride (over- the- counter type of vitamin B6) 200 mg po bid
  Arms: pyridoxamine
Drug: placebo — placebo
  Arms: identical placebo

SUMMARY:
The purpose of this study is to determine if a specific form of Vitamin B known as Pyridoxamine helps improve bone strength over one year in women (>65 yrs old) with Type 2 Diabetes. The investigators know that people with type 2 diabetes have the lower bone material strength and the investigators suspect this is due to high levels of circulating sugars that build up over time (known as Advanced Glycation Endproducts). The investigators will study whether using a specific form of vitamin B, known as pyridoxamine helps improve bone strength and reduce levels of circulating sugars over a one year time period.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) has become one of the most important diseases of our time. Recent research shows that diabetes has negative effects on bones and that people with diabetes might more likely to break a bone. The investigators don't know the reasons for this, but the investigators suspect that normal bone replacement is slowed down in diabetes and this could slow down the growth of new bone. It is possible that the normal material becomes weaker because sugar-related components ("Advanced Glycation Endproducts") are making the bone more brittle. The investigators have shown in past research that people who have type 2 diabetes are more likely to have both weaker bone with lower "bone material strength" and also higher level of sugar-related components("Advanced Glycation Endproducts"). This study will focus on attempting to lower the sugar-related components("Advanced Glycation Endproducts") by treating a group of patients with type 2 diabetes with an over- the- counter B vitamin, known as vitamin B6 or pyridoxamine for one year. The investigators will compare post-menopausal women both before and after pyridoxamine use and study them in terms of different bone features based on blood tests, bone imaging, a bone indentation test and a measurement of sugar-related components in the skin. This study will help to clarify if using pyridoxamine helps improve bone strength in women with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women ≥65 years
* Diagnosis of T2D for ≥ 5 years, with all HbA1c levels.

Exclusion Criteria:

* Hormone replacement treatment (HTR) use (to avoid the influence of estrogen).
* Fractures (excluding skull, facial bones, metacarpals, fingers, toes, and fractures associated with severe trauma) within 12 months.
* A history of pathological fractures (eg, due to Paget's disease, myeloma, metastatic malignancy).
* Type 1 diabetes
* Disorders associated with altered skeletal structure or function (chronic liver disease' chronic renal disease stage 4 [eGFR < 30 mL/mim/1.73 m2] or worse, malignancy, hypoparathyroidism or hyperparathyroidism,acromegaly, Cushing's syndrome, hypopituitarism, alcohol intake > 3U/day).
* Treatment with any of the following drugs in part year:current corticosteroid, anticonvulsant therapy(phenytoin, phenobarbital, primidone, carbamazepine), SGLT2 inhibitor if on it for < 1 year), pharmacological doses of thyroid hormone (TSH<normal), adrenal or anabolic steroids, Aromatase inhibitors, calcitonin, bisphosphonates, denosumab, estrogen, or selective estrogen receptor modulator, sodium fluoride, teriparatide, thiazolidinediones(TZDs).
* Serum 25(OH)D levels < 20 ng/ml. If 25(OH)D levels are < 20 ng/ml, rescreening will be allowed following a vitamin D loading regimen of 50,000 IU/week for 4 weeks. If serum 25(OH) D levels are ≥ 20 ng/ml after supplementation, the subject will be allowed to enroll.
* Current use of pyridoxamine (although not multivitamin or vitamin B6 users because pyridoxamine is not at pharmacologic levels in these supplements).
* Allergy to pyridoxamine and vitamin B6.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Bone formation in serum by P1NP | 12 months
  change in serum biochemical marker of bone formation, P1NP

SECONDARY OUTCOMES:
Advanced glycation endproducts | 12 months
  Skin assessment of advanced glycation endproducts

CONTACTS AND LOCATIONS:
Overall Officials: Mishaela Rubin,, M.D, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - Harkness Pavillion, New York, New York, United States

DOCUMENTS (1):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT03778580/Prot_000.pdf